CLINICAL TRIAL: NCT02696343
Title: Somatosensory Modulation of Salivary Gene Expression and Oral Feeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Tufts Medical Center (Other); CIRI/CHI Institute for Research and Innovation (Unknown); California Institute for Medical Research (Other); Texas Tech University (Other); Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UNL IRB Project ID #15446
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Infant, Extremely Low Birth Weight; Feeding Behavior
Keywords: somatosensory stimulation; orocutaneous; gene expression
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPI experimental (Experimental): Preterm infants randomized to receive the PULSED orocutaneous somatosensory stimulation from the NTrainer during tube feedings.
  Interventions: Device: NTrainer
- EPI control (Sham Comparator): Preterm infants randomized to receive the Sham (blind pacifier) during tube feedings.
  Interventions: Device: SHAM blind pacifier

INTERVENTIONS:
Device: NTrainer — pulsed orocutaneous stimulation paired with tube feedings
  Arms: EPI experimental
Device: SHAM blind pacifier — regular green Soothie pacifier paired with tube feedings
  Arms: EPI control

SUMMARY:
Two innovative approaches, pulsatile orocutaneous entrainment of non-nutritive suck via orosensory entrainment (NTrainer) device technology and serial salivary gene expression analyses, will be merged to examine the relation between gene expression, oral somatosensory stimulation, feeding behavior, and neurodevelopmental outcomes at 18 months corrected age (CA) on 180 extremely preterm infants [EPIs] (24 0/7-26 6/7 GA and 27 0/7 - 28 6/7 GA) enrolled at three neonatal intensive care units: Catholic Health Initiative (CHI) Health St. Elizabeth (Lincoln, NE), Tufts Medical Center (Boston, MA), and Santa Clara Valley Medical Center (San Jose, CA). EPIs will be randomized to a blind pacifier (SHAM) or PULSED NTrainer treatment groups, and stratified by GA, sex, and bronchopulmonary dysplasia status (BPD vs non-BPD). We hypothesize that the combination of the NTrainer® intervention for improved oral feeding skills, along with objective salivary gene expression data to monitor response to treatment and feeding development, will result in a novel, objective, and personalized approach to neonatal oral feeding and reduce the duration of time to attain oral feeds while improving feeding, growth and neurodevelopmental outcomes at 18 months' CA.

DETAILED DESCRIPTION:
The purpose of this study is to combine molecular and behavioral methods in an experimental conceptualization approach to map the effects of trigeminal (PULSED orocutaneous) somatosensory stimulation on salivary gene expression in the context of the acquisition of an exquisitely complex oromotor skill, namely oral feeding, in high-risk human neonates. The aims of this study represent the first attempt to combine non-invasive treatment strategies and transcriptomic assessments of high-risk EPIs to (1) improve oral feeding behavior and skills, (2) further our understanding of the gene ontology of biologically diverse pathways related to oral feeding, (3) use gene expression data to personalize neonatal care and individualize treatment strategies and timing interventions, and (4) improve long-term developmental outcomes. This integrative approach to oral feeding is a paradigm shift in neonatal care where rapidly emerging technological advances and personalized transcriptomics can safely and non-invasively be brought to the neonatal bedside to inform medical care decisions and improve care and outcomes.

Methods Participants: Only EPIs born between 24 0/7 and 28 6/7 weeks' gestation, as determined by obstetric ultrasound at < 15 weeks or last menstrual period, are eligible to participate in this study. We will actively enroll EPIs once they have a corrected PCA of ≥ 29 weeks to limit the number of infants who develop serious sequelae of prematurity and would not be eligible for this study based upon the criteria listed below. Parents of enrolled subjects will receive a Babies R Us $50 gift card for their participation. Subjects will be recruited from four neonatal intensive care units including 1) CHI Health St. Elizabeth [Lincoln, NE], 2) Tufts Medical Center NICU [Boston, MA], 3) Santa Clara Valley Medical Center [San Jose, CA], and 4) Childrens Hospital Orange Country [Los Angeles, CA] by a study site PI/Co-Investigator or the neonatal study coordinator. Informed consent will be obtained prior to participants' entry into the study, following consultation with the attending physician and nurse(s). A total of 180 EPIs (approximately equal numbers of males and females, no exclusion based on race/ethnicity) will participate in the study (power >.85, Type I error <.05).

Exclusion criteria: EPIs will not be recruited for this study if they have any of the following: 1) chromosomal and congenital anomalies including craniofacial malformation, nervous system anomalies, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia and/or other major gastrointestinal anomalies; 2) congenital infection, 3) no documented GA, 4) severe IUGR (3%), 5) abnormal neurological status including head circumference < 10th or > 90th percentile, intracranial hemorrhage grades III and IV, seizures, meningitis, neurological examination showing abnormal tone or movements of all extremities for PCA; 6) history of necrotizing enterocolitis (stage II and III); and, 7) culture-positive sepsis at the time of study enrollment.

Protocol: EPIs will be stratified among two gestational age groups (24 0/7 - 26 6/7 weeks, and 27 0/7 - 28 6/7 weeks). Each infant will be randomized to receive either the PULSED NTrainer or SHAM intervention using a software random integer function in Minitab v.17 (www.minitab.com). Infants assigned to the PULSED NTrainer group will receive a progressive dose of the pulsatile orocutaneous stimulation. Beginning at 30 weeks' PCA, these infants will receive 2 weeks of low-dose PULSED NTrainer stimulation (2 x 3-minute blocks) with a 1-minute stimulus 'off-period' between the stimulation blocks. This form of stimulation will be given simultaneous with tube feedings 3 times/day. The stimulus dose will then be increased over the next 2 weeks (3 x 3-minute blocks of PULSED NTrainer stimulation) with a 1-minute stimulus 'off-period' between the stimulation blocks, also given simultaneously with tube feedings 3 times/day. EPIs randomized to the SHAM condition will be given a regular silicone pacifier during tube feedings over the same time period.

A 1-minute rest period (no stimulation) occurs between stimulation blocks. Criteria for initiation of orocutaneous therapy include the following: 1) stable vital signs and not on continuous vasopressor medications; 2) tolerating enteral feeds in previous 48 hours; and 3) not intubated and mechanically ventilated. If the infant is on nasal intermittent positive pressure ventilation, continuous positive airway pressure or nasal cannula >2 liters per minute, then the FiO2 must be <40%.

NNS Assessment and Automated NNS Digital Signal Processing and Feature Extraction: In addition to the oral stimulation interventions (PULSED NTrainer vs. SHAM pacifier), all study infants will be assessed 3 times/week (e.g., M/W/F) for NNS performance. The NTrainer System will be used in 'assessment mode' to record the compression dynamics of NNS during a 3-minute session to immediately precede a tube feeding that is not associated with an intervention condition.

The most active 2-minute period of NNS behavior based on suck cycle count is automatically extracted from each suck assessment data file using an automated waveform feature extraction algorithm on the NTrainer System. Pressure peaks > 1.6 cm H2O are subjected to feature extraction criteria, including suck cycle symmetry, cycle duration, and burst identification defined as two or more NNS events occurring within 1200 ms. This algorithm permits objective identification of NNS burst activity distinct from non-NNS mouthing compressions or tongue thrusts against the pacifier. Four measures will be objectively extracted from the indexed records of suck compression, including minute-rates for (1) NNS Bursts where an individual burst includes 2 or more suck cycles, (2) NNS Cycle Events defined as suck compression cycles with cycle periods less than 1200 ms, (3) Total Oral Compressions defined as the sum of all pressure events, and (4) NNS compression pressure expressed in cm H2O.

PO Feeding Advancement: EPIs will advance on a standardized cue-based feeding schedule utilized by each site NICU, known as Infant Driven Feeding® that will lead to full nipple feeds. This standardization of oral feeding advancements across sites will limit confounders that may ultimately skew the data.

Saliva Collection, Processing, and Gene Expression Analysis: Saliva Collection: Saliva samples will be collected from all enrolled infants on the first day prior to receiving either the SHAM or PULSED NTrainer intervention. This sample will serve as our baseline gene expression profile. Samples will then be obtained twice per week (~ 3 day intervals) up to the time of achievement of full oral feeds or discharge home from the hospital with either a nasogastric tube (NG) or gastronomy tube.

Saliva samples at each site will be collected with techniques that have been optimized and validated through the Maron laboratory. Briefly, saliva samples will be collected with a 1 mL syringe, end caps removed and attached to low wall suction. Saliva will be collected for approximately 20 seconds and immediately stabilized in 500 μL of Qiagen's RNA Protect Saliva to halt gene expression changes, inhibit destructive RNases, and limit microbial overgrowth. Samples will be vortexed briefly and frozen at -20 deg C. Once frozen, samples are stable for up to 18 months prior to the need for total RNA extraction. Thus, samples from Nebraska and Santa Clara will be shipped once a month on ice overnight to the Maron laboratory at the Mother Infant Research Institute at Tufts Medical Center in Boston, MA for processing.

Generation of a Saliva Biobank: One additional saliva sample will be obtained each week from all enrolled subjects to generate a biobank repository. Banking an additional sample each week from study subjects will ensure that we will limit loss of data points. We anticipate that there are informative salivary biomarkers of oral feeding maturation that have yet to be identified. By generating a biobank of additional saliva samples that may be retrospectively interrogated on either a microarray gene expression platform or with RNASeq, we will have the potential to discover novel hypotheses about gene-gene interactions and/or transcriptional regulatory processes related to oral feeding in the EPI population.

Total RNA Extraction: Salivary samples will extracted for total RNA using established protocols optimized in the Maron laboratory. RNA extraction will occur with the QIAGEN RNAProtect Saliva Mini kit per manufacturer's instructions. On column DNase treatment will be performed for each sample to eliminate genomic DNA contamination. Samples that are part of the biobank will be frozen at -80°C pending need for future analysis. Samples that will be used for RT-qPCR experiments will first undergo cDNA conversion with the Life Technologies SuperScript Vilo kit per manufacturer's instructions. cDNA will be stored at -80°C in the Mother Infant Research Institute at Tufts Medical Center pending gene expression analysis.

Gene Expression Analysis: For the purpose of this study, we will interrogate each sample for nine genes, six target genes of interest and three reference genes for quality control and potential normalization of gene expression data. Genes to be analyzed in this study have been previously shown to be directly linked to oral feeding in the newborn and include PLXNA1, PLXNA3, NPY2R, WNT3, AMPK, and NPHP4. The three reference genes include GAPDH, HPRT1, and YWHAZ, all of which have been shown to maintain stable gene expression across advancing PCA. All cDNA samples will undergo a targeted pre-amplification with a custom TaqMan® PreAmp Master Mix for all nine genes. This targeted approach to amplification will ensure that only those genes of interest will be amplified and not all genes across the transcriptome which may introduce bias. Preamplified cDNA will then undergo PCR with TaqMan Fast Advance Master Mix on the Life Technologies Quant Studio 7 Flex Real-Time PCR System. This instrument is housed with the Mother Infant Research Institute at Tufts Medical Center and is an advanced state-of-the-art PCR machine and software system. All efforts will be made to adhere to the Minimum Information for Publication of Quantitative Real-Time PCR Experiments (MIQE) guidelines for this study. All samples will be run in duplicate with appropriate positive and negative controls.

Initial Gene Expression Analyses: All gene expression data will be normalized on the Quant Studio 7 Flex Real-Time PCR System. Only samples that have successful amplification of all three reference genes will be considered in the analysis. Previously, genes have been informative in a binary fashion (+/- expression). However, for the purpose of this study, we will be prepared to calculate relative gene expression of each target gene with the delta delta cycle threshold (ΔΔCt) method. In accordance to the MIQE guidelines, we will use the three reference genes for normalization and determine a geometric mean of their Ct in each sample to calculate relative gene expression.

Neurodevelopmental Follow-Up: As part of standard of care, each site will complete the Bayley Scales of Infant and Toddler Development 3rd Edition, on EPIs at 18 to 24 months' corrected age (CA). The primary subtests of interest include Fine Motor, Gross Motor, Cognition, and Language. These data will be recorded, analyzed, and correlated with feeding outcomes in the neo-and post-natal period, gene expression data, and intervention status. In addition, growth parameters including head circumference, length and weight will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants (EPIs) born between 24 0/7 and 28 6/7 weeks' GA, as determined by obstetric ultrasound at < 15 weeks or last menstrual period
* Enroll EPIs once they have a corrected PCA of ≥ 29 weeks
* Approximately equal numbers of males and females, no exclusion based on race/ethnicity

Exclusion Criteria:

* Chromosomal and congenital anomalies including craniofacial malformation, nervous system anomalies, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia and/or other major gastrointestinal anomalies
* Congenital infection
* No documented GA
* Severe IUGR (3%)
* Head circumference < 10th or > 90th percentile
* Intracranial hemorrhage grades III and IV, seizures
* Meningitis
* Neurological examination showing abnormal tone or movements of all extremities for PCA
* History of necrotizing enterocolitis (stage II and III)
* Culture-positive sepsis at the time of study enrollment

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Salivary gene expression | Quantify gene expression probability from salivary samples beginning at 30 wks post-menstrual age, and repeated sampling every 3 days thereafter during the infant's stay in neonatal intensive care unit (NICU) for an average of 14 samples, up to 60 days.
  Plexin A1 (PLXNA1), Plexin A3 (PLXNA3), Neuropeptide Y2 receptor (NPY2R), Wingless-type integration site family (WNT3), Adenosine-monophosphate-activated protein kinase (AMPK), and Nephronophthisis 4 (NPHP4) gene expression

SECONDARY OUTCOMES:
National Institute Child Human Development (NICHD) Neonatal Research Network feed-growth questionnaire | 18 months corrected age (CA)
  Growth and feeding progression and mode of feeding following NICU discharge up to 18 months
Bayley III Developmental Scales | 18-24 months corrected age (CA)
  Assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior
Non-nutritive suck (NNS) bursts/minute | Beginning at 30 wks post-menstrual age, and repeated biomechanical sampling of suck bursts/min (2 min sample) every 3 days thereafter during the infant's stay in the NICU for an average of 12 NNS samples, and up to 60 days.
  NNS Bursts/min
Time-to-transition to full oral feed | Time expressed in days for an infant to attain full oral feed (100% PO), assessed on a daily basis beginning at 30 weeks post-menstrual age (PMA) through hospital stay in the NICU, for an average of 56 %PO measures sampled over 8 weeks.
  Time to Full Oral Feed
Non-nutritive suck cycles/min | Beginning at 30 wks post-menstrual age, and repeated biomechanical sampling of suck compressions/min (2-min sample) every 3 days thereafter during the infant's stay in the NICU for an average of 12 NNS samples, and up to 60 days.
  NNS Cycles/min
Non-nutritive suck Spatiotemporal Index (NNS STI) | Beginning at 30 wks post-menstrual age, and repeated biomechanical sampling of suck compressions/min (2-min sample) every 3 days thereafter during the infant's stay in the NICU for an average of 12 NNS samples, and up to 60 days.
  NNS STI based on 5 suck bursts and the first 5 suck compression cycles
Non-nutritive suck compression amplitude (cmH2O) | Beginning at 30 wks post-menstrual age, and repeated biomechanical sampling of suck compressions/min (2-min sample) every 3 days thereafter during the infant's stay in the NICU for an average of 12 NNS samples, and up to 60 days.
  NeoNNS.exe batch measure of peak suck pressure during NNS burst production

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Barlow, PhD, Principal Investigator — University of Nebraska; Jill L Maron, MD, Principal Investigator — Tufts Medical Center
Locations (4):
- United States (4):
  - Children's Hospital of Orange County, Los Angeles, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Tufts Medical Center, Boston, Massachusetts
  - CHI St. Elizabeth's Medical Center, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Barlow SM, Maron JL, Alterovitz G, Song D, Wilson BJ, Jegatheesan P, Govindaswami B, Lee J, Rosner AO. Somatosensory Modulation of Salivary Gene Expression and Oral Feeding in Preterm Infants: Randomized Controlled Trial. JMIR Res Protoc. 2017 Jun 14;6(6):e113. doi: 10.2196/resprot.7712. PMID 28615158